CLINICAL TRIAL: NCT01243736
Title: Assessment of Combined Bowel Preparation for Capsule Endoscopy Study
Acronym: CEPREP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Stephanie L. Hansel, Assistant Professor of Medicine, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 10-000198
Record Dates: First submitted 2010-10-19; First posted 2010-11-18 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Gastrointestinal Hemorrhage
Keywords: anemic; bleeding; blood in stool; abdomen pain; Gastrointestinal bleeding; capsule endoscopy (CE)
MeSH Terms: conditions — Gastrointestinal Hemorrhage; Hemorrhage; Abdominal Pain | interventions — Polyethylene Glycols; Simethicone; Metoclopramide

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard prep (No Intervention): One group will receive the standard bowel preparation, which consists of eating no solid foods after 7 p.m. the evening prior to the capsule endoscopy test and being able to consume clear liquids up to 4 hours prior to the capsule endoscopy test
- Combination Prep (Active Comparator): The other group will receive the combination bowel preparation, which consists of taking the standard bowel preparation plus:
  1. drinking 2-liters (8 cups) of polyethylene glycol starting at 7 p.m. the night prior to the capsule endoscopy test;
  2. drinking a teaspoon of simethicone 20 minutes prior to the capsule endoscopy test;
  3. drinking a teaspoon of metoclopramide 20 minutes prior to the capsule endoscopy test;
  4. lying on your right side for 30 minutes following the swallowing of the capsule endoscope.
  Interventions: Drug: Combination Prep

INTERVENTIONS:
Drug: Combination Prep — combination bowel preparation, which consists of:
  1. drinking 2-liters (8 cups) of polyethylene glycol starting at 7 p.m. the night prior to the capsule endoscopy test;
  2. drinking a teaspoon of simethicone 20 minutes prior to the capsule endoscopy test;
  3. drinking a teaspoon of metoclopramide 20 minutes prior to the capsule endoscopy test;
  4. lying on your right side for 30 minutes following the swallowing of the capsule endoscope.
  Other Names: polyethylene glycol; simethicone; metoclopramide
  Arms: Combination Prep

SUMMARY:
The investigators are conducting a study to see if taking a bowel preparation before having a capsule endoscopy is more helpful than the standard preparation of not eating after 7 PM the night before a capsule endoscopy in making it easier to see the small bowel in order to find the source of gastrointestinal bleeding.

DETAILED DESCRIPTION:
This is a single-blind, prospective randomized controlled study to determine if a combination of purgative agent, prokinetic agent, simethicone, and position will improve small bowel visualization, diagnostic yield, and completion rate of capsule endoscopy.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years old
2. Gastrointestinal bleeding as indication for capsule endoscopy.
3. Ability to give informed consent

Exclusion Criteria:

1. Subject has an allergy to polyethylene glycol or other adverse reaction to a previous bowel preparation with PEG3350 (MoviPrep®), metoclopramide, or simethicone;
2. Subjects has gastrointestinal motility disorder;
3. Subjects had stomach or small bowel resection;
4. Pregnancy;
5. Subjects has pheochromocytoma;
6. Subjects has uncontrolled hypertension;
7. Subjects has seizure disorders;
8. Subjects has concurrent MAO inhibitor use;
9. Subject has G6PD deficiency;
10. Subjects has swallowing disorder (including impaired gag reflex);
11. Subjects has hyponatremia with serum sodium less than 130 mm0l/L

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-04; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Improvement small bowel visualization, diagnostic yield, and complete rate of capsule endoscopy | 1 year
  The primary endpoints of small bowel visualization quality, diagnostic yield, and completion rate will be compared between groups using Pearson's chi-square test.

SECONDARY OUTCOMES:
Safety outcomes and Patient satisfaction | 1 year
  secondary endpoints of safety outcomes and patient satisfaction with Pearson's chi-square test.
gastric transit time | 1 year
  A group comparison for the secondary outcome of gastric transit time will be done using a two-sample t-test or Wilcoxon rank-sum test, as appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie L. Hansel, M.D., Principal Investigator — Mayo Clinic; Elizabeth Rajan, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Hansel SL, Murray JA, Alexander JA, Bruining DH, Larson MV, Mangan TF, Dierkhising RA, Almazar AE, Rajan E. Evaluating a combined bowel preparation for small-bowel capsule endoscopy: a prospective randomized-controlled study. Gastroenterol Rep (Oxf). 2019 Oct 19;8(1):31-35. doi: 10.1093/gastro/goz054. eCollection 2020 Feb. PMID 32419949